CLINICAL TRIAL: NCT02432378
Title: A PHASE 2 EFFICACY TRIAL OF INTENSIVE LOCOREGIONAL CHEMOIMMUNOTHERAPY FOR ADVANCED STAGE OVARIAN CANCER AND TUMOR-SPECIFIC INTRANODAL AUTOLOGOUS ALPHA-DC1 VACCINES
Brief Title: Intensive Locoregional Chemoimmunotherapy for Recurrent Ovarian Cancer Plus Intranodal DC Vaccines
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: AIM ImmunoTech Inc. (Industry); National Cancer Institute (NCI) (NIH); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCI 11-128/IC 3050822; 5P01CA132714 (NIH)
Record Dates: First submitted 2015-04-08; First posted 2015-05-04 (Estimated); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Cancer of Ovary; Cancer of the Ovary; Neoplasms, Ovarian; Ovarian Cancer; Ovary Cancer; Ovary Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Cisplatin; Celecoxib; Creatine Kinase, MM Form

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cisplatin + Celecoxib + DC Vaccine (Experimental): Cisplatin 50 mg/m2 by IP once per cycle (21 days) + celecoxib daily 200 mg by mouth daily + intranodal vaccine injections once per cycle
  Interventions: Biological: Cisplatin + celecoxib + DC vaccine
- Cisplatin + CKM + Celecoxib + DC Vaccine (Experimental): Cisplatin 50 mg/m2 by IP once per cycle (21 days) + celecoxib daily 200 mg by mouth daily + IFN by IP once per cycle + rintatolimod 200 mg by IP once per cycle + intranodal vaccine injections once per cycle
  Interventions: Biological: Cisplatin + CKM + Celecoxib + DC Vaccine

INTERVENTIONS:
Biological: Cisplatin + celecoxib + DC vaccine — Cisplatin 50 mg/m2 by IP once per cycle (21 days) + celecoxib daily 200 mg by mouth daily + intranodal vaccine injections once per cycle
  Arms: Cisplatin + Celecoxib + DC Vaccine
Biological: Cisplatin + CKM + Celecoxib + DC Vaccine — Cisplatin 50 mg/m2 by IP once per cycle (21 days) + celecoxib daily 200 mg by mouth daily + IFN by IP once per cycle + rintatolimod 200 mg by IP once per cycle + intranodal vaccine injections once per cycle
  Arms: Cisplatin + CKM + Celecoxib + DC Vaccine

SUMMARY:
This study will evaluate the immunologic and potential clinical effectiveness of intensive locoregional sequential intraperitoneal (IP) cisplatin (IPC) with intravenous (iv) paclitaxel followed by peritoneal infusion of a chemokine modulatory (CKM) regimen composed of a cocktail of IP rintatolimod and interferon-alpha (IFNα) for patients with advanced stage ovarian cancer (III-IV) at primary neoadjuvant setting.

In the safety phase I phase, we determined the tolerable dose of IPC-CKM. In this phase 2 we will add intradermal (ID) autologous αDC1 vaccines (known to be nontoxic) to the tolerable IPC-CKM regimen. The effectiveness will be determined by rate of complete pathologic response.

DETAILED DESCRIPTION:
On Phase 1, patients received up to 6 cycles of IPC, with CKM after the 2nd to 6th cycles. On Phase 2, (which opened 8/27/24/ )patients will receive up to 6 -8 cycles of chemotherapy with ID injections of DC1 vaccine with CKM. To optimize the pattern of immunity, all patients will also receive oral celecoxib (COX2 inhibitor).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have advanced stage (III-IV) epithelial carcinoma of ovarian, tubal, or peritoneal origin.

  * Histologic documentation of the original primary tumor is required via the pathology report.
  * Original tumor blocks from primary diagnosis biopsy will be reviewed by our study pathologist at Magee.
  * Patients must be receiving neoadjuvant chemotherapy
* Patients must be eligible for cancer-related definitive therapy with neoadjuvant chemotherapy
* Patients must be chemonaive and receiving therapy in primary first line neoadjuvant setting
* Patients must have GOG performance of 0-1
* Patients must be reasonable candidates for interval debulking surgery as well as IP platinum based combination chemotherapy regimen with no prior evidence of clinically significant intra-abdominal adhesions, persistent abdominal wall infections, renal toxicity, or bowel obstruction.
* Patients of childbearing potential must have a negative pregnancy test prior to the study entry and be practicing an effective form of contraception. If applicable, patients must discontinue breastfeeding prior to the first date of treatment on this study.
* Patient must be willing to undergo leukapheresis
* Patients must agree to appropriate clinical monitoring to receive the study regimens.
* Patient must have:

  * Bone marrow function:
  * Absolute neutrophil count (ANC) greater than or equal to 1,500/µL, equivalent to CTCAE v4 grade 1.
  * Platelets greater than or equal to 100,000/µL;
  * hemoglobin greater than or equal to 8.0 g/dL.
* Renal function:

  * creatinine less than or equal to 1.5 x institutional upper limit normal (ULN), CTCAE v4 grade 1.
* Hepatic function:

  * Bilirubin less than or equal to 1.5 x ULN (CTCAE v4 grade 1).
  * SGOT and alkaline phosphatase less than or equal to 2.5 x ULN (CTCAE v4 grade 1).
* Patients who have signed informed consent and authorization permitting release of personal health information.
* Patients must have a GOG Performance Status of 0 or 1.
* Exclusion Criteria:
* Patients who have an active autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus (SLE), ulcerative colitis, Crohn's Disease, multiple sclerosis (MS), ankylosing spondylitis).
* Patients with a known allergy to cisplatin or taxane chemotherapy. Patients with carboplatin allergy may be included if they tolerate a test dose of IV cisplatin given in monitored floor conditions. Patients who are allergic to paclitaxel, can be alternatively treated with abraxane.
* Patients being chronically treated with immunosuppressive drugs such as cyclosporin, adrenocorticotropic hormone (ACTH), or systemic corticosteroids.
* Patients with a recognized immunodeficiency disease including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia; patients who have acquired, hereditary, or congenital immunodeficiencies.
* Patients with uncontrolled diseases other than cancer will be excluded.
* Patients who are pregnant or nursing.
* Patients who have contraindications to the use of NSAID's like chronic renal failure, coronary artery disease, or bleeding ulcers.
* Patients with tumors of low malignant potential, except ovarian pseudomyxoma or with no peritoneal disease.
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.
* Patients with previous pelvic radiation therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-09-04 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Change in the number of CD8+ tumor infiltrating T cells in the peritoneal fluid. | 8 weeks
  The difference in CD8+ tumor infiltrating T cells over 3 cycles of platinum based chemotherapy plus immunotherapy compared with baseline.
Number of adverse events for the different combinations | 8 weeks
  2 patients will be treated and observed for 2 cycles on each of the dose tiers to identify the acceptable dose of IFN in combination with the other protocol drugs/vaccine for the second phase of the trial.

SECONDARY OUTCOMES:
Change in the number of CD3+CD8+ T cells in the peritoneal fluid. | 8 weeks
Change in the number of effector CD8+ T cells in the peritoneal fluid. | 8 weeks
Change in the number of CD4+ T cells in the peritoneal fluid. | 8 weeks
Change in the number of Tregs in the peritoneal fluid. | 8 weeks
Change in the number of myeloid-derived suppressor cells in the peritoneal fluid. | 8 weeks

OTHER OUTCOMES:
Change in the number of TH1 cells in the peritoneal fluid. | 8 weeks
Change in the number of natural killer cells in the peritoneal fluid. | 8 weeks
Change in the number of dendritic cells in the peritoneal fluid. | 8 weeks
Change in the number of activated macrophages in the peritoneal fluid. | 8 weeks
Change in the number of tumor cells in the peritoneal fluid. | 8 weeks
Change in the concentration of CCL3 in the peritoneal fluid. | 8 weeks
Change in the concentration of CCL4 in the peritoneal fluid. | 8 weeks
Change in the concentration of CCL5 in the peritoneal fluid. | 8 weeks
Change in the concentration of CXCL9 in the peritoneal fluid. | 8 weeks
Change in the concentration of CXCL10 in the peritoneal fluid. | 8 weeks
Change in the concentration of CXCL11 in the peritoneal fluid. | 8 weeks
Change in the concentration of CXCL12 in the peritoneal fluid. | 8 weeks
Change in the concentration of GrB in the peritoneal fluid. | 8 weeks
Change in the concentration of IFN gamma in the peritoneal fluid. | 8 weeks
Change in the concentration of FoxP3 in the peritoneal fluid. | 8 weeks
Change in the concentration of IDO in the peritoneal fluid. | 8 weeks
Change in the concentration of NO in the peritoneal fluid. | 8 weeks
Change in the concentration of IL-10 in the peritoneal fluid. | 8 weeks
Change in the concentration of COX-2 in the peritoneal fluid. | 8 weeks
Change in the number of CD3+ cells in the tumor tissue. | 8 weeks
Change in the number of CD4+ cells in the tumor tissue. | 8 weeks
Change in the number of CD8+ cells in the tumor tissue. | 8 weeks
Change in the number of CD11b+ cells in the tumor tissue. | 8 weeks
Change in the number of CD11c+ cells in the tumor tissue. | 8 weeks
Change in the number of GrB+ cells in the tumor tissue. | 8 weeks
Change in the number of FoxP3+ cells in the tumor tissue. | 8 weeks
Change in the number of IDO+ cells in the tumor tissue. | 8 weeks
Change in the number of CCL3 cells in the tumor tissue. | 8 weeks
Change in the number of CCL4 cells in the tumor tissue. | 8 weeks
Change in the number of CCL5 cells in the tumor tissue. | 8 weeks
Change in the number of CXCL9 cells in the tumor tissue. | 8 weeks
Change in the number of CXCL10 cells in the tumor tissue. | 8 weeks
Change in the number of CXCL11 cells in the tumor tissue. | 8 weeks
Change in the number of CCL22 cells in the tumor tissue. | 8 weeks
Change in the number of CXCL12 cells in the tumor tissue. | 8 weeks
Change in the number of GrB cells in the tumor tissue. | 8 weeks
Change in the number of IFN gamma cells in the tumor tissue. | 8 weeks
Change in the number of FoxP3 cells in the tumor tissue. | 8 weeks
Change in the number of IDO cells in the tumor tissue. | 8 weeks
Change in the number of NO cells in the tumor tissue. | 8 weeks
Change in the number of IL-10 cells in the tumor tissue. | 8 weeks
Change in the number of COX-2 cells in the tumor tissue. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Edwards, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC CancerCenter at Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Hillman Cancer Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Orr B, Mahdi H, Fang Y, Strange M, Uygun I, Rana M, Zhang L, Suarez Mora A, Pusateri A, Elishaev E, Kang C, Tseng G, Gooding W, Edwards RP, Kalinski P, Vlad AM. Phase I Trial Combining Chemokine-Targeting with Loco-Regional Chemoimmunotherapy for Recurrent, Platinum-Sensitive Ovarian Cancer Shows Induction of CXCR3 Ligands and Markers of Type 1 Immunity. Clin Cancer Res. 2022 May 13;28(10):2038-2049. doi: 10.1158/1078-0432.CCR-21-3659. PMID 35046055